CLINICAL TRIAL: NCT00669396
Title: A Pilot Study of Copper T380A IUDs Versus Oral Levonorgestrel for Emergency Contraception
Brief Title: Copper T380 IUD Versus Oral Levonorgestrel for Emergency Contraception vs. Plan B for Emergency Contraception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Turok, PI, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23111; IUDvsPlanBforEC
Record Dates: First submitted 2008-04-25; First posted 2008-04-30 (Estimated); Results first posted 2009-08-06 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Pregnancy
Keywords: contraception; emergency contraception; pregnancy prevention after unprotected intercourse
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): IUD
  Interventions: Drug: Copper T380 IUD
- 2 (Active Comparator): Oral levonorgestrel
  Interventions: Drug: levonorgestrel

INTERVENTIONS:
Drug: Copper T380 IUD — Copper T380 IUD
  Other Names: Paragard IUD
  Arms: 1
Drug: levonorgestrel — 1.5 mg
  Other Names: Plan B
  Arms: 2

SUMMARY:
The purpose of this study is to see if women presenting for emergency contraception (EC) are willing to accept the copper intrauterine device (IUD). This study will also compare the use of effective methods of contraception between women who selected the copper IUD or Plan B 6 months after they received EC.

DETAILED DESCRIPTION:
This study seeks to estimate the acceptance of Copper IUD use amongst people presenting for EC. This will be accomplished by offering all women who present for EC at participating Planned Parenthood Association of Utah (PPAU) clinics during the study period the option of having the copper IUD or Plan B. Women who agree to study participation will be followed for 6 months. The primary outcome for the study is the use of a reliable method of contraception 6 months after presenting for EC.

Secondary outcomes measured will be pregnancies, abortions, repeat Plan B use, presence of gonorrhea or Chlamydia infection at the time of presentation for EC, number of days to first bleeding episode and duration of that bleeding episode, further bleeding patterns, frequency of unprotected intercourse, use of a barrier method for prevention of sexually transmitted infections, patient satisfaction with the chosen method and symptoms possibly related to contraception use. Patients selecting the IUD will be assessed for IUD expulsion, perforation, and removal.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-45 years old, in need of EC (had unprotected intercourse within 120 hours), willing to give consent for participation in research, willing to comply with the study requirements, and accessible by telephone.
* Patients selecting the IUD need to identify themselves as desiring long-term contraception.

Exclusion Criteria:

* Current pregnancy,
* Had pelvic inflammatory disease or a septic abortion within the past 3 months or gonorrheal or chlamydial infection in the last 60 days,
* Current behavior suggesting a high risk for pelvic inflammatory disease
* Allergy to copper, or Wilson's disease (for patients selecting Paragard) or allergy to levonorgestrel (for patients selecting Plan B)
* Intracavitary of symptomatic uterine fibroids, and abnormalities of the uterus that distort the uterine cavity,
* Mucopurulent cervicitis,
* A previously placed IUD that has not been removed
* Genital bleeding of unknown etiology
* Ovarian, cervical or endometrial cancer,
* Small uterine cavity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD/MPH, Principal Investigator — University of Utah
Locations (1):
- Planned Parenthood Association of Utah, West Valley City Clinic, West Valley City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Copper T380 IUD: IUD
- Levonorgestrel: Oral levonorgestrel
Period: Overall Study
Arm/Group | Copper T380 IUD | Levonorgestrel
Started | 23 | 34
Completed | 13 | 22
Not Completed | 10 | 12
Not completed — Lost to Follow-up | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Copper T380 IUD | Levonorgestrel | Total
Number analyzed (Participants) | 23 | 34 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 34 | 57
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (6.7) | 23.0 (4.7) | 23.7 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 34 | 57
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 34 | 57

OUTCOME MEASURES:

1. Primary Outcome: Use of an Effective Method of Contraception at 6 Months After Requesting Emergency Contraception
Description: Use of a method of contraception with a typical efficacy rate >= to 92%. This includes combined hormonal contraception (combined oral contraceptive pills, the contraceptive patch and ring), sterilization, IUDs, Depo-provera, and contraceptive implants.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Copper T380 IUD | Levonorgestrel
Number analyzed (Participants) | 13 | 22
participants | 9 | 13

2. Secondary Outcome: Pregnancy
Description: positive urine pregnancy test at anytime within 6 months of presenting for emergency contraception.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Copper T380 IUD | Levonorgestrel
Number analyzed (Participants) | 13 | 22
participants | 0 | 2

3. Secondary Outcome: Infection
Description: diagnosis and treatment for pelvic inflammatory disease
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Copper T380 IUD | Levonorgestrel
Number analyzed (Participants) | 13 | 22
participants | 0 | 0

4. Secondary Outcome: IUD Expulsion, Removal, or Perforation
Description: patient reports IUD expulsion, removal, or perforation OR one of these events was documented at the clinic where patient received care.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Copper T380 IUD | Levonorgestrel
Number analyzed (Participants) | 13 | 22
participants | 5 | 0

ADVERSE EVENTS:
Arm/Group | Copper T380 IUD | Levonorgestrel
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/34
Other Adverse Events (participants affected / at risk) | 0/23 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No